CLINICAL TRIAL: NCT00195845
Title: A Phase 4 Double-Blind, Placebo-Controlled Study of Galantamine to Improve Cognitive Dysfunction in Bipolar Disorder
Brief Title: A Double-Blind, Placebo-Controlled Study of Galantamine to Improve Cognitive Dysfunction in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHA-IRB-0000/02/03; GAL-USA-T102
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double-Blind Galantamine vs Placebo (Experimental): Double-Blinded, Placebo-Controlled Study of Galantamine to Improve Cognitive Dysfunction
  Interventions: Drug: Galantamine
- Placebo Control Group (Placebo Comparator): Placebo-Controlled Group
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Galantamine
  Arms: Double-Blind Galantamine vs Placebo
Drug: Placebos
  Arms: Placebo Control Group

SUMMARY:
The purpose of this study is to determine if galantamine augmentaion improves cognition in euthymic bipolar patients. In addition, the effect of galantamine on clinical measures of functioning and psychopathology will also be assessed.

DETAILED DESCRIPTION:
The study length is 12 to 24 weeks depending on whether patients enter the crossover. Study also involves 3 neuropsychology testings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60; DSM-IV diagnosis of bipolar disorder, any subtype; Baseline Mini Mental Status exam above 20; MRS < 16; MADRS < 16

Exclusion Criteria:

* Current substance dependence; serious unstable medical conditions; active suicidal ideation; current DSM-IV for a major mood episodes; history of COPD, epilepsy, cardiac arrhythmia, and peptic ulcer disease; meet DSM-IV criteria for dementia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Primary Completion 2006-09 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Dunn, MD, PhD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States